CLINICAL TRIAL: NCT03672110
Title: Slow and Low Start of a Tacrolimus Once Daily Immunosuppressive Regimen: A Multicentre Prospective Randomized Controlled Study
Brief Title: Slow and Low Start of a Tacrolimus Once Daily Immunosuppressive Regimen
Acronym: S&L
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-SplusL-061
Record Dates: First submitted 2014-10-08; First posted 2018-09-14 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Renal Failure; Renal Insufficiency; Renal Disease; Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Renal Insufficiency, Chronic

ARMS (2):
- Standard tacrolimus group (Active Comparator): Control group: Advagraf will be administered as usual (0.2mg/kg bodyweight), trough levels will be measured every day in the first week after kidney transplantation (TX) and Advagraf dose will be adjusted accordingly.
  Interventions: Drug: Advagraf
- Fixed dose tacrolimus group (Experimental): Study group: Advagraf will be administered per fix dose 5mg/day, trough levels will be blinded during the first week, there will be no adjustments in the first week after TX.
  Interventions: Drug: Advagraf

INTERVENTIONS:
Drug: Advagraf — intervention: different advagraf dosing in the study compared to the control arm, see above
  Other Names: no other intervention name

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of an advagraf based immunosuppressive regimen with slower dose tapering and lower starting dose of Advagraf compared with a standard Advagraf-based immunosuppressive regimen in de novo renal transplantation. Non inferiority will be assessed by a combined study endpoint consisting of the development of biopsy-proven rejection of BANFF class Ia or higher and/or graft loss and/or patient death within the first six months after renal transplantation.

DETAILED DESCRIPTION:
The most widely used immunosuppressive regimen, in adult kidney transplant recipients, consists of an induction therapy accompanied by maintenance with tacrolimus, mycophenolate and steroids. In the long term, tacrolimus is the single most effective immunosuppressive agent. For adult kidney transplant recipients maintenance of therapeutic levels remains crucial regarding the prevention of allograft rejections. Greater blood levels variability is associated with inferior graft survival as well as non-adherence. Lower variability of tacrolimus blood levels after conversion to extended release tacrolimus formulations has been shown. In addition, once-daily administration promotes patient adherence. The latter is one of the major causes for allograft loss.

In the first week after kidney transplantation stable tacrolimus blood levels are hardly achievable. Especially extended release tacrolimus formulations often yield high tacrolimus blood levels. High blood levels are a known risk factor for delayed graft function, which leads to a prolonged hospitalization and a reduced graft survival. Additionally high blood levels are associated with polyomavirus infections and may increase the incidence of new-onset diabetes after renal transplantation.

Taking this into consideration, authors demand for calcineurin inhibitor (CNI)-free immunosuppression or the delayed onset of CNI therapy after a stable graft function is reached. This would inevitably lead to a higher rate of acute allograft rejections in the early phase after kidney transplantation. Avoiding high tacrolimus levels, especially early after transplantation, to minimize delayed graft function as well as long term undesirable side effects, seems particularly necessary.

For early dose adjustments of extended release tacrolimus formulations, more medical experience is needed compared to immediate release formulations. More stable tacrolimus blood levels can be seen after the first week of administration.

To avoid high blood levels of tacrolimus, especially early after transplantation, the investigators aim to demonstrate in this study a non-inferiority of a low dose extended release tacrolimus regimen compared to a standard extended release tacrolimus-based immunosuppressive regimen in de novo renal transplantation. Given inclusion criteria and excluding the exclusion criteria, participants will be randomized into two groups, a standard tacrolimus administration group with daily dose adjustments within the first week after transplantation and a fixed dose tacrolimus administration group, without dose adjustments within the first week after transplantation. In the first 6 months after renal transplantation different blood levels of tacrolimus shall be reached. In the case of the standard tacrolimus administration group the investigators aim at tacrolimus blood levels of 7-9 ng/ml in the first 2 months after transplantation and 6-8 ng/ml for days 61 to 180. In the fixed dose tacrolimus administration group, the low extended release tacrolimus dose of 5mg per day well no be changed in the first week after transplantation. For safety reasons blinded measurements will take place in the first week and study officials will be alerted in case of repeated tacrolimus levels > 20 ng/ml. On days 7 to 60 the investigators aim at tacrolimus blood levels of 5-7 ng/ml and from days 61 to 180 4-6 ng/ml. Non inferiority will be assessed by a combined study endpoint consisting of the development of biopsy-proven rejection of BANFF class Ia or higher and/or graft loss and/or patient death within the first six months after renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* male or female allograft recipients at least 18 years old
* primary or secondary kidney transplantation
* deceased or living donor
* normal immunological risk profile (PRA level > 20%, AB0-compatible donation, negative crossmatch)
* informed consent of the patient

Exclusion Criteria:

* graft loss due to severe rejection within the first year after transplantation (in case of secondary transplantation)
* multi-organ recipient
* patients receiving a kidney from a non-beating donor
* complete human leukocyte antigen (HLA)-identical living donor (twins)
* patients with a history of malignancy during the last five years (except squamous or basal cell carcinoma of the skin after successful treatment)
* patients with uncontrolled infectious disease, particularly patients who are HIV-positive or suffer from chronic hepatitis B or C or tuberculosis
* patients with severe gastroenteric disorder, particularly severe diarrhea and symptoms of enteric malabsorption
* patients suffering from liver cirrhosis CHILD B or C or other severe liver disease (aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), GammaGT ≥ 3-fold increased)
* thrombopenia < 70,000/mm3
* leukopenia < 2,500/mm3
* participation in another clinical trial within the last 4 weeks prior to inclusion
* estimated addiction or other disorders that do not allow the person concerned, the nature and scope and possible consequences of the clinical trial
* pregnant or breast-feeding women
* women of childbearing age, except women who meet any of the following criteria: post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum > 40 U/ml, postoperatively (6 weeks after bilateral oophorectomy with or without hysterectomy), regular and correct use of a contraceptive method with error rate < 1 % per year (e. g. implants, depot injections, oral contraceptives, intrauterine device IUD), sexual abstinence, vasectomy of the partner
* evidence that the patient is likely to fail to comply with the protocol (e. g. lack of cooperation)
* hypersensitivity to Advagraf or a product listed in the prescribing information other component as well as to other macrolides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-09; Primary Completion 2020-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint: defined as biopsy-proven acute rejection, graft loss or death between the groups at month 6 post-transplantation in renal transplantation) | 6 months after transplantation
  combined endpoint: defined as biopsy-proven acute rejection, graft loss or death between the groups at month 6 post-transplantation in renal transplantation

SECONDARY OUTCOMES:
Rate of necessary dose modifications to achieve Advagraf target levels in early post-op period | 6 months after transplantation
  rate of necessary dose modifications in order to achieve Advagraf target levels in the early postoperative period
Improved renal transplant function in the early postoperative period and 6 months post-op | 6 months after transplantation
  renal function defined by need for renal replacement therapy as well as by means of glomerular filtration rate
Lower incidence of delayed graft function (DGF) | 6 months after transplantation
  rate of DGF defined as need for at least one postoperative hemodialysis
Reduced incidence of new onset diabetes after renal Transplantation (NODAT) | 6 months after transplantation
  incidence of NODAT. Diabetes mellitus defined by American Diabetes Association - Guidelines 2016
Reduced rates of infection | 6 months after transplantation
  incidence of viral or other infections
Incidence of malignancies | 6 months after transplantation
  incidence rate of biopsy proven malignancies
Incidence of fractures | 6 months after transplantation
  incidence rate of radiography or clinically proven fractures
Incidence of heart failure | 6 months after transplantation
  incidence rate of heart failure
Incidence of myocardial infarction | 6 months after transplantation
  incidence rate of myocardial infarction
Incidence of venous thrombosis | 6 months after transplantation
  incidence rate of venous thrombosis proven by color-coded duplex sonography or radiography
Incidence of peripheral vascular disease | 6 months after transplantation
  incidence rate of peripheral vascular disease, sonography or radiography proven
Incidence of cerebrovascular disease | 6 months after transplantation
  incidence rate of cerebrovascular disease, sonography or radiography proven
Incidence of hypercholesterolemia | 6 months after transplantation
  hypercholesterolemia is defined as > upper limit of normal and measured in mmol/L
Incidence of hypertriglyceridemia | 6 months after transplantation
  hypertriglyceridemia is defined as > upper limit of normal and measured in mmol/L
Incidence of hyperlipoproteinemia | 6 months after transplantation
  hyperlipoproteinemia is defined as low density lipoproteins cholesterol > upper limit of normal and measured in mmol/L
Incidence of hypolipoproteinemia | 6 months after transplantation
  hypolipoproteinemia is defined as high density lipoproteins cholesterol < lower limit of normal and measured in mmol/L
Incidence of dyslipidemia | 6 months after transplantation
  dyslipidemia is defined as low density lipoproteins cholesterol > upper limit of normal and high density lipoproteins cholesterol < lower limit of normal and each measured in mmol/L
Incidence of arterial hypertension | 6 months after transplantation
  blood pressure is measured in mm of mercury (mmHg) and arterial hypertension is defined according to the American College of Cardiology 2017 Guideline for High Blood Pressure in Adults
Incidence of anemia | 6 months after transplantation
  anemia is defined as hemoglobin level or erythrocyte count < lower limit of normal and measured in mmol/L or Tpt/L respective
Incidence of cardiovascular mortality | 6 months after transplantation
  cardiovascular mortality is defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident
Chronic humoral rejection | 6 months after transplantation
  Rate of biopsy proven chronic humoral rejections
Interstitial fibrosis and tubular atrophy as histological changes in renal transplant biopsies | 6 months after transplantation
  interstitial fibrosis and tubular atrophy are expressed as percentage in biopsy reports
Incidence of polyomavirus nephropathy | 6 months after transplantation
  polyomavirus nephropathy is defined by simian virus 40 (SV40) positive histological staining in renal transplant biopsies
Recurrence rate of the underlying kidney disease requiring renal transplantation | 6 months after transplantation
  Biopsy proven recurrence of the underlying disease
Rate of donor-specific antibodies | 6 months after transplantation
  rate of donor-specific antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hugo, MD, PhD, Principal Investigator — TU Dresden
Locations (1):
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany